CLINICAL TRIAL: NCT01283113
Title: Evaluation of Intra-Abdominal Fat Contents in Patients With Type 2 Diabetes Using a Novel Non-Invasive Method of Bioelectric Impedance
Brief Title: Evaluation of Intra-Abdominal Fat in Patients With Type 2 Diabetes Using a Non-Invasive Method
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Osama Hamdy, Principal Investigator, Joslin Diabetes Center
Other Study IDs: CHS # 2010-01
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Type 2 Diabetes; Metabolic Syndrome
Keywords: Visceral Fat; Waist Circumference; Bioelectrical Impedance; Metabolic Syndrome; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of this study is to compare 2 different measurements of visceral fat that can be easily used in clinical practice (waist circumference versus bioelectric impedance) in relation to known risk factors of coronary artery disease in a large cohort of patients with type 2 diabetes and with a BMI range between 20-45 kg/m2

ELIGIBILITY:
Inclusion Criteria:

* Established type 2 diabetes
* Age 18 - 80
* Body mass index (BMI) between 20-45 Kg/m2.
* Willing to undergo laboratory and anthropometric assessments.

Exclusion Criteria:

* The study will not include women who are pregnant, or are not using reliable birth control methods or who they think that they might be pregnant due to potential risk of fetal affection.
* Subjects with known malignancy, treated or untreated will be excluded (except treated skin melanoma).
* Subjects with major psychological problems or a major eating disorder will be excluded.
* Subjects with heart Pacemaker or any other electronic devices attached to their body will be excluded.
* Subjects with confirmed type 1 diabetes or positive anti GAD antibodies test will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will identify and recruit 500 patients. Participants for this study (men and women) will be recruited for the diabetes outpatient clinic of the Joslin Diabetes Center. Subjects from minority and various ethnic/racial groups will be invited to participate in the study at the same proportional to Massachusetts's population, which is 86.5% white, 6.9 Black, 0.3% American Indian and Alaska, 4.9 Asian, 0.1% Native Hawaiian and Other Pacific Islander and 8.2% of Hispanic or Latino origin. The investigators will monitor our recruitment by gender and race/ethnicity and modify our recruitment procedures if necessary to ensure that there is no selection bias due to these factors.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Visceral fat level | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, M.D., Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States